CLINICAL TRIAL: NCT01518673
Title: National Study of Low Dose Effects of X-rays in Pediatric Patients Undergoing a CT Examination.
Brief Title: Low Dose Effects of X-rays in Pediatric Patients Undergoing a CT Examination.
Acronym: PedCTBe
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Federal Agency for Nuclear Control, Belgium (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2010/708
Record Dates: First submitted 2012-01-20; First posted 2012-01-26 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Pediatric Patients Undergoing a Computed Tomography Examination
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood lymphocytes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- X-rays
  Interventions: Procedure: Blood test

INTERVENTIONS:
Procedure: Blood test — Analysing X-ray induced genetic effects in pediatric patients directly after a computer tomography scan.

SUMMARY:
Patients undergoing a computed tomography are exposed to a relatively high dose of X-rays. Pediatric patients are known to be very radiosensitive with respect to radiation induced cancer. Using the technique of scoring γ-H2AX foci in peripheral blood lymphocytes the most important lesions to the genetic material DNA, double strand breaks induced by CT X-rays can be detected. The technique will be applied in a multicenter setting for evaluation of X-effects induced by a computed tomography examination in a population of pediatric patients. To this end a blood sample will be taken from the patients before and after the examination.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients wearing a catheter

Exclusion Criteria:

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients undergoing computed tomography are exposed to a relatively high dose of X-rays.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
X-ray induced genetic effects in pediatric patients directly after a computed tomography scan. | Within 30 min after the computed tomography examination.
  Assessment of γ -H2AX foci in peripheral blood lymphocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Smeets, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be